CLINICAL TRIAL: NCT01946802
Title: Trial of Device for Seizure Detection Using SEDline During Therapeutic Hypothermia in Cardiac Arrest Victims
Brief Title: Seizure Detection Using SEDline During Therapeutic Hypothermia in Cardiac Arrest Victims
Status: Completed | Type: Observational
Sponsor: Gil Joon Suh (Other)
Collaborators: Masimo Corporation (Industry); Humed Co., Ltd (Unknown)
Responsible Party: Sponsor-Investigator, Gil Joon Suh, Professor, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Other Study IDs: H-1303-013-470
Record Dates: First submitted 2013-09-11; First posted 2013-09-20 (Estimated); Results first posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Cardiac Arrest
Keywords: Heart arrest; Cardiopulmonary resuscitation; Hypothermia induced; Seizures; Electroencephalography
MeSH Terms: conditions — Heart Arrest; Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Frontal 4 channel EEG: Consecutive comatose patients admitted to the emergency ICU for postresuscitation care following successful cardiopulmonary resuscitation after nontraumatic out-of-hospital and in-hospital cardiac arrest.
  Interventions: Device: Frontal 4 channel EEG

INTERVENTIONS:
Device: Frontal 4 channel EEG — Simultaneous conventional EEG and SEDline monitoring for 30 minutes during and after therapeutic hypothermia
  Other Names: SEDline, Masimo corporation

SUMMARY:
Current guidelines recommend the use of sedatives and neuromuscular blocking agents to avoid shivering during therapeutic hypothermia in cardiac arrest victims. Therefore, it is difficult to detect seizure and the frequent or continuous EEG monitoring is recommended. However, it is difficult to follow this recommendation in most clinical situations due to the lack of specialized devices and persons. The purpose of this study is whether SEDline (frontal 4-channel EEG device) has a diagnostic value to detect seizure during therapeutic hypothermia in cardiac arrest victims.

DETAILED DESCRIPTION:
1. Treatment of cardiac arrest victims Enrolled patients receive basic and advanced cardiac life support according to the 2010 American Heart Association (AHA) Guidelines for Cardiopulmonary Resuscitation (CPR) and Emergency Cardiovascular Care (ECC).

   After acquiring sustained return of spontaneous circulation (ROSC), the patients are immediately admitted to the ICU and are provided postresuscitation care including mild therapeutic hypothermia for 24 hours post-ROSC.

   During therapeutic hypothermia, their core temperatures are maintained from 32 to 34°C.

   Then rewarming is conducted (< 0.25°C/hour) till core temperature 36.5°C. To avoid shivering, we use sedatives and neuromuscular blocking agents during the therapeutic hypothermia.
2. Conventional EEG Conventional EEG is conducted for 30 minutes at

   1) During therapeutic hypothermia and rewarming (within 72 hours after cardiac arrest) Then, the results are interpreted by a neurologist for the presence of seizure.
3. SEDline SEDline is monitored during the simultaneous period with the conventional EEG. Data retrieved from the SEDline are blindly interpreted by 3 investigators to determine the presence of seizure activity.

   The presence of seizure activity in SEDline is determined by the definition
   1. Electrographic seizure: rhythmic discharge or spike and wave pattern with definite evolution in frequency, location, or morphology lasting several seconds.
   2. Spike: Transient, clearly distinguishable from background activity, with pointed peak at conventional paper speeds and a duration of 20 to less than 70 ms
4. Anti-epileptic drug The use of anti-epileptic drugs is guided by the results of conventional EEG or the presence of clinically seizure-like movement
5. Gold standard The presence of Seizure identified in conventional EEG.
6. Primary outcome The diagnostic performance of SEDline to detect seizure will be tested: Sensitivity, specificity, positive predictive value, negative predictive value, accuracy, and area under receiver operating characteristics curve (AUC).

ELIGIBILITY:
Inclusion Criteria:

* Consecutive comatose patients admitted to the emergency ICU for postresuscitation care following successful cardiopulmonary resuscitation after nontraumatic out-of-hospital and in-hospital cardiac arrest.
* Cardiac arrest is defined as cessation of cardiac mechanical activity, confirmed by the absence of a detectable pulse, unresponsiveness, and apnea.

Exclusion Criteria:

* Age < 18 years old
* Contraindication to therapeutic hypothermia: active life-threatening bleeding, septic shock, or refractory fatal arrhythmia..
* Intracranial pathology including hemorrhage or tumor
* Visible generalized seizure before the study enrollment
* Advanced directives to withdraw life-sustaining treatment
* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Comatose cardiac arrest survivors admitted to a 12-bed emergency intensive care unit of Seoul National University Hospital, Seoul, Republic of Korea.
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2014-12; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gil Joon Suh, Prof, Study Director — Seoul National University Hospital
Locations (1):
- Department of Emergency Medicine, Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
After discussion with Masimo

REFERENCES:
- [Background] HOCKADAY JM, POTTS F, EPSTEIN E, BONAZZI A, SCHWAB RS. ELECTROENCEPHALOGRAPHIC CHANGES IN ACUTE CEREBRAL ANOXIA FROM CARDIAC OR RESPIRATORY ARREST. Electroencephalogr Clin Neurophysiol. 1965 May;18:575-86. doi: 10.1016/0013-4694(65)90075-1. No abstract available. PMID 14296835
- [Background] Rossetti AO, Urbano LA, Delodder F, Kaplan PW, Oddo M. Prognostic value of continuous EEG monitoring during therapeutic hypothermia after cardiac arrest. Crit Care. 2010;14(5):R173. doi: 10.1186/cc9276. Epub 2010 Sep 29. PMID 20920227
- [Background] Crepeau AZ, Rabinstein AA, Fugate JE, Mandrekar J, Wijdicks EF, White RD, Britton JW. Continuous EEG in therapeutic hypothermia after cardiac arrest: prognostic and clinical value. Neurology. 2013 Jan 22;80(4):339-44. doi: 10.1212/WNL.0b013e31827f089d. Epub 2013 Jan 2. PMID 23284064

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Form 31/12/2014 to 19/08/2016 In the Emergency Intensive Care Unit of Seoul National University Hospital
Pre-assignment Details: 53 were screened for eligibility. 9 were excluded (4 Advanced directives to withhold or withdraw life-sustaining treatment, 3 No informed consent, 1 Known intracranial pathology, and 1 Visible generalized seizure). 44 provided informed consents. 5 were withdrawn(see baseline characteristics). Finally 39 patients were enrolled.
Groups:
- Frontal 4 Channel EEG: Consecutive comatose patients admitted to the emergency ICU for postresuscitation care following successful cardiopulmonary resuscitation after nontraumatic cardiac arrest.
Period: Overall Study
Arm/Group | Frontal 4 Channel EEG
Started | 44
Completed | 39
Not Completed | 5
Not completed — Death | 1
Not completed — Withdrawal by Subject | 2
Not completed — Combined septic shock | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: 44 provided informed consents. Among them 5 were withdrawn. 1 death before EEG, 2 relative withdrew patient, 1 combined septic shock, and 1 patient did not perform EEG within 72 hours.
  Finally 39 patients were enrolled in this study.
Arm/Group | Frontal 4 Channel EEG
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 18
Age, Continuous [Median (Full Range); unit: years] | 60 [34 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 25
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 39

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Seizure-positive and Seizure-negative That Were Correctly Classified by the SEDline in All Evaluated Cases
Description: Conventional EEG (gold standard for seizure detection) and SEDline monitoring will be conducted simultaneously for 30 minutes at During therapeutic hypothermia and rewarming (12 ~ 72 hours after cardiac arrest). Then, data retrieved from the conventional EEG and SEDline will be interpreted and analyzed for the presence of seizure.
Time Frame: Within 72 hours after cardiac arrest
Population: 44 provided informed consents. Among them 5 were withdrawn. 1 death before EEG, 2 relative withdrew patient, 1 combined septic shock, and 1 patient did not perform EEG within 72 hours.
  Finally 39 patients were enrolled in this study. Conventional EEG (gold standard for seizure detection) and SEDline monitoring were conducted simultaneously for 30 minutes at During therapeutic hypothermia and rewarming.
Measure: Number; unit: percentage of seizures
Arm/Group | Frontal 4 Channel EEG
Number analyzed (Participants) | 39
percentage of seizures | 100

2. Secondary Outcome: Sensitivity of SEDline for Seizure Detection
Description: Sensitivity measured the percentage of seizures identified by the SEDline in cases those were identified as seizures by the conventional EEG.
Time Frame: Within 72 hours after cardiac arrest
Measure: Number; unit: percentage of seizure (+)
Arm/Group | Frontal 4 Channel EEG
Number analyzed (Participants) | 39
percentage of seizure (+) | 100

3. Secondary Outcome: Specificity
Description: Specificity measured the percentage of seizure-negative identified by the SEDline in cases those were identified as seizure-negative by the conventional EEG.
Time Frame: Within 72 hours after cardiac arrest
Measure: Number; unit: percentage of seizure (-)
Arm/Group | Frontal 4 Channel EEG
Number analyzed (Participants) | 39
percentage of seizure (-) | 100

4. Secondary Outcome: Positive Predictive Value
Description: Positive predictive value measured the percentage of seizures identified by the conventional EEG in cases those were identified as seizures by the SEDline.
Time Frame: Within 72 hours after cardiac arrest
Measure: Number; unit: percentage of seizure (+)
Arm/Group | Frontal 4 Channel EEG
Number analyzed (Participants) | 39
percentage of seizure (+) | 100

5. Secondary Outcome: Negative Predictive Value
Description: Negative predictive value measured the percentage of seizure-negative identified by the conventional EEG in cases those were identified as seizure-negative by the SEDline.
Time Frame: Within 72 hours after cardiac arrest
Measure: Number; unit: percentage of seizure (-)
Arm/Group | Frontal 4 Channel EEG
Number analyzed (Participants) | 39
percentage of seizure (-) | 100

6. Secondary Outcome: Area Under Receiver Operating Characteristics Curve (AUC) of SEDline for Seizure Detection
Description: The Area under receiver operating characteristics curve (AUC) of SEDline represents the accuracy of the SEDline to detect seizures compared with the conventional EEG.
Time Frame: Within 72 hours after cardiac arrest
Measure: Number; unit: probability
Arm/Group | Frontal 4 Channel EEG
Number analyzed (Participants) | 39
probability | 1.00

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Frontal 4 Channel EEG
All-Cause Mortality (participants affected / at risk) | 17/39
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 0/39

LIMITATIONS AND CAVEATS:
Since the SEDline system provides 4-channel-processed EEG monitoring in the frontal area, focal seizures could not be detected and spatial localization of the seizure might be difficult.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes